CLINICAL TRIAL: NCT06930911
Title: Analysis of Antibiotic Stewardship to Prevent Early Sepsis in Infants Less Than 35 Weeks of Age, With a View to Its Optimization
Brief Title: Antibiotic Stewardship to Prevent Early Sepsis in Preterm Infants
Acronym: BACTINEO
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 25-5057
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Prematurity, Infections
MeSH Terms: conditions — Premature Birth; Infections | interventions — Anti-Infective Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Preterm infant: Patients born before 35 weeks and admitted in the tertiary neonatal unit of the Croix Rousse between 01/01/2021 and 31/12/2023.
  Interventions: Biological: Antibiotic therapy

INTERVENTIONS:
Biological: Antibiotic therapy — Evaluating antibiotic exposure in premature infants before 35 weeks in a tertiary care neonatal unit

SUMMARY:
Early onset sepsis (EOS) occurs in newborns within the first 72 hours of life, and is rare, about 0.8 cases per 1000 births (1). It is more frequent in premature infants and potentially more severe (as much as 75% of deaths has been reported in extreme premature infants (1)). Infection is considered as confirmed when blood or cerebral fluid cultures detect a pathogen (1). It is considered probable when cultures are negative, but there are clinical (fever, hemodynamic failure, severe respiratory condition) and biological (inflammatory markers) signs suggestive of infection. In 2017, French recommendations for prevention of EOS in term and near-term infants has been proposed. However, to date, there are no recommendations for the population of premature newborns, and there are discrepancies in practices antibiotic stewardship to prevent early sepsis in infants born before 35 weeks. Preterm infants are more exposed to EOS than infants born closer to term. The incidence is inversely proportional to gestational age, reaching 32 cases per 1000 births in infants born between 22 and 24 weeks. Infection is a major cause of mortality and morbidity in premature newborns, because of the immaturity of their immune system. The death rate reach 50% in infants born between 22 and 28 weeks. For these reasons, probabilistic antibiotic therapy is prescribed at admission in Neonatology in 35 to 50% of very premature babies. But it appears that the prescription of antibiotics is not correlated with the incidence of EOS, with overuse of antibiotics, related to the fear of infection in these fragile patients. However, exposure to antibiotics induces gut dysbiosis, which is the main risk factor of necrotizing enterocolitis, a potentially severe disease occurring specifically in preterm infants. It is therefore important to optimize antibiotic stewardship in the days following birth, to improve the quality of care. To this end, we shall analyse antibiotic prescription practices and the rate of EOS in premature newborns hospitalized in a tertiary care unit at the Croix Rousse university hospital.

ELIGIBILITY:
Inclusion Criteria:

* - infants born at a gestational age of less than 35 weeks - Born between January 1, 2021 and December 31, 2023

Exclusion Criteria:

* - Parent refusal

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Infants born before 35 weeks hospitalized in neonatology at croix rousse hospital.
Sampling Method: Probability Sample
Enrollment: 711 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of premature infants treated with antibiotics | During the first three days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Croix Rousse hospital, Lyon, France